CLINICAL TRIAL: NCT03089697
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase IIa Clinical Study to Evaluate Safety and to Explore Efficacy of N-Rephasin® SAL200, in Patients With Persistent Staphylococcus Aureus Bacteremia
Brief Title: Phase IIa Clinical Study of N-Rephasin® SAL200
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment into this study was terminated by the Sponsor prior to completion for strategic reasons.
Sponsor: Intron Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITB-101
Record Dates: First submitted 2017-02-23; First posted 2017-03-24 (Actual); Results first posted 2021-08-17 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Staphylococcus Aureus Bacteremia; Anti-Bacterial Agents
Keywords: N-Rephasin SAL200; Methicillin-Sensitive Staphylococcus aureus; Methicillin Resistant Staphylococcus Aureus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-Rephasin® SAL200 (Experimental): To assign the study group, administer the conventional standard treatment (CST) (antibiotics) for MRSA/MSSA with N-Rephasin® SAL200 (3mg/kg); N-Rephasin® SAL 200 is given by intravenous only once at Day 1.
  Interventions: Biological: N-Rephasin® SAL200
- Placebo (Placebo Comparator): To assign the control group, administer the conventional standard treatment (CST) (antibiotics) for MRSA/MSSA with Formulation buffer (placebo); Placebo (INT200) is given by intravenous only once at Day 1 (same way with Experimental group)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: N-Rephasin® SAL200 — A single dose of SAL200 (SAL-1, 3mg/kg) intravenous administration of the study drug, in addition to the conventional standard treatment (antibiotics) for MRSA/MSSA
  Arms: N-Rephasin® SAL200
Other: Placebo — A single dose of the formulation buffer (placebo), excluding the main ingredient of the study drug in addition to the conventional standard treatment (antibiotics) for MRSA/MSSA
  Arms: Placebo

SUMMARY:
This study is performed to evaluate safety and to explore the efficacy of a single intravenous dose of N-Rephasin® SAL200 (3 mg/kg) in addition to the conventional standard treatment, for persistent Staphylococcus aureus bacteremia in patients, for more than 48 hours even after antibiotic treatment to which Staphylococcus aureus is susceptible.

DETAILED DESCRIPTION:
Subjects:

Patients with persistent Staphylococcus aureus bacteremia for more than 48 hours from the beginning of antibiotics treatment to which Staphylococcus aureus is susceptible.

Study Method:

1. Selection of patients with persistent S.aureus bacteremia for more than 48 hours even after application of the standard treatment for S. aureus bacteremia
2. Randomization according to the trial institutions
3. The control group receives a single intravenous dose of the placebo in addition to the standard treatment for persistent Staphylococcus aureus bacteremia
4. The study group receives a single intravenous dose of the N-Rephasin® SAL200 (3 mg/kg) in addition to the standard treatment for persistent Staphylococcus aureus bacteremia
5. A blood culture is performed 18 hours (±6 hours) after the administration of N-Rephasin® SAL200
6. Blood cultures continue to be performed every 24 hours (±6 hours) or 48 hours (±6 hours) after the previous blood culture, until two consecutive results of 'no growth (negative conversion)' are obtained
7. Adverse events are monitored at the time of the first blood culture following the administration of N-Rephasin® SAL200 or placebo, and at the subsequent intervals of 24 hours or 48 hours

Statistical Analysis:

1. Primary endpoints

   * Safety analysis is conducted in the Safety group. A distribution table of patients who experience at least one adverse event (incidence), and distribution tables of the relationship of the reported adverse events with the investigational product (distribution tables for severity and the relationship with the drug) are presented with respect to the groups (study group, control group), to determine safety of the investigational product.
   * The results of the laboratory tests, anaphylaxis test, inflammatory cytokine test and vital signs at baseline and the last visit are summarized as mean values and standard deviations, to determine the change before and after the treatment within each group.
   * Categorical data are divided into normal and abnormal, and summarized as the frequency and percentage to determine the difference before and after treatment within each group.
2. Secondary endpoints

   * Proportion of patients who are negative for bacterial growth in the first blood culture after administration of the investigational drug. The descriptive statistics for the proportion of patients who are negative for bacterial growth in the first blood culture (the rate of no growth) after the first treatment are presented by treatment group. Whether the rate of no growth is superior in the study group compared to the control group, is evaluated by a descriptive statistical method.
   * Proportion of patients who die due to S. aureus bacteremia by Day14 after the incidence of bacteremia. The descriptive statistics for the proportion of patients who die due to S. aureus bacteremia by Day14 are presented by treatment group and evaluated.
   * Proportion of treatment failure for S. aureus bacteremia by Day 14 (if two consecutive results of 'no growth' are not achieved in the blood cultures which are performed until Day 14. The descriptive statistics for the proportion of treatment failure for S. aureus bacteremia by Day 14 are presented and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MSSA/MRSA bacteremia who are confirmed to have more than a pair of Gram positive bacteria in a blood culture conducted at 48~96 hours after the start of antibiotic treatment to which S. aureus is susceptible.
2. Males or females aged 19 years or older
3. Those who understand the explanatory notes for subjects, and sign the informed consent.

Exclusion Criteria:

1. Those who do not receive appropriate antibiotics within 48 hours after the occurrence of bacteremia (the time point of reporting it to the department of laboratory medicine)
2. The Gram positive strain, identified in a blood culture conducted at 48~96 hours after the start of antibiotic treatment to which S. aureus is susceptible, is not the same strain of S. aureus which was cultured when the definite diagnosis of S. aureus bacteremia was made
3. Those who pass 48 hours after confirmation of persistent S. aureus bacteremia through a blood culture conducted at 48~96 hours after the start of antibiotic treatment to which S. aureus is susceptible
4. Those who have symptoms of septic shock at the time of acquisition of the consent form

   * Systolic blood pressure lower than 90 mmHg, or blood pressure lower than usual by more than 40 mmHg, in spite of the application of appropriate fluid therapy
   * Requirement of hypertensor to maintain the systolic blood pressure at 90 mmHg or higher
5. Those who were infected with mixed bacterial species
6. Those who are hypersensitive to N-Rephasin® SAL200, who have a clinically significant hypersensitivity to it, or a past history there of
7. Pregnant or lactating women and women of child-bearing potential (who do not agree to take appropriate contraceptive measures during the trial period)
8. Those who participated in other clinical trial within 30 days prior to enrollment
9. Patients with any conditions that may interfere with study participation or accurate evaluation on investigator's judgment
10. Those who may die within 72 hours due to other serious complications (e.g., cerebral infarction, etc.), as per the investigator's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Bin Kim, M.D, PhD, Principal Investigator — Seoul National University Bundang Hospital; Wan Beom Park, M.D, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kundsin RB. Documentation of airborne infection during surgery. Ann N Y Acad Sci. 1980;353:255-61. doi: 10.1111/j.1749-6632.1980.tb18928.x. No abstract available. PMID 6939390
- [Result] Etienne J, Fleurette J, Ninet JF, Favet P, Gruer LD. Staphylococcal endocarditis after dental extraction. Lancet. 1986 Aug 30;2(8505):511-2. doi: 10.1016/s0140-6736(86)90377-6. No abstract available. PMID 2875256
- [Result] Lamy B, Dargere S, Arendrup MC, Parienti JJ, Tattevin P. How to Optimize the Use of Blood Cultures for the Diagnosis of Bloodstream Infections? A State-of-the Art. Front Microbiol. 2016 May 12;7:697. doi: 10.3389/fmicb.2016.00697. eCollection 2016. PMID 27242721
- [Result] van Hal SJ, Jensen SO, Vaska VL, Espedido BA, Paterson DL, Gosbell IB. Predictors of mortality in Staphylococcus aureus Bacteremia. Clin Microbiol Rev. 2012 Apr;25(2):362-86. doi: 10.1128/CMR.05022-11. PMID 22491776
- See also: Frency J, Brun Y, Bes M, Meugnier H, Grimont F, Grimon PAD, Newi C, Fleurette J. Staphylococcus lugdunensis sp. and Staphylococcus schleiferi sp. novel two species from human clinical specimens. Int Syst Bacteriol. 1998;38:168-172 — https://www.microbiologyresearch.org/content/journal/ijsem/10.1099/00207713-38-2-168
- See also: Seung-Ho Han et al., Monitoring of Methicillin-Resistant Staphylococcus aureus in Nasal Swabs Obtained fron Dental Clinic Healthcare Providers and Medical Environments Nurses. Int J Oral Biology. 2010;35:7-12 — https://www.kci.go.kr/kciportal/ci/sereArticleSearch/ciSereArtiView.kci?sereArticleSearchBean.artiId=ART001432619
- See also: Hyuk Min Lee, Dong Eun Yong, Kyungwon Lee., Antimicrobial Resistance of Clinically Important Bacteria Isolated from 12 Hospitals in Korea in 2004 . Korean Journal of Clinical Microbiology 2005;8(1):66-73 — https://ir.ymlib.yonsei.ac.kr/handle/22282913/147505
- See also: Woo J-H, Song J-H, Cheong H-S, Lee E-K, Chae S-M, Kim N-J. Analysis of Economic Outcomes of Methicillin-Resistant Staphylococcus Aureus(MRSA) Bacteremia Using Retrospective Case-Control Study. Korean J Clin Pharm 2007;17(2):59-64. — http://www.ekjcp.org/journal/view.html?uid=329&sort=&scale=&key=year&keyword=&s_v=17&s_n=2&pn=vol&year=2007&vmd=Full
- See also: Lee, H, Yong, D, Lee, K, Hong, S, Kim, E, Jung, S, Park, Y, Choi, T, Eo, Y, Shin, J et al. Antimicrobial Resistance of Clinically Important Bacteria Isolated from 12 Hospitals in Korea in 2004. Korean J Clinical Microbiology 2005;8(1):66-73 — https://www.koreamed.org/SearchBasic.php?RID=2224695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | N-Rephasin® SAL200
Started | 13 | 12
Completed | 11 | 10
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | N-Rephasin® SAL200 | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Full Range); unit: Years] | 64.23 [36.0 to 88] | 65.33 [34.0 to 93.0] | 64.8 [34.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 13 | 12 | 25
Height (cm) [Mean (Full Range); unit: cm] | 165.19 [144.90 to 186.00] | 161.96 [148.00 to 175.00] | 163.6 [144.90 to 186.00]
Weight (kg) [Mean (Full Range); unit: kg] | 60.35 [43.90 to 79.30] | 59.03 [40.40 to 71.40] | 59.7 [40.40 to 79.30]

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoints - Summary of Treatment-emergent Adverse Events (Safety Set)
Description: The safety analysis was conducted based on the data of all AEs, physical examinations, clinical laboratory tests, and vital signs (blood pressure, pulse rate, body temperature, and respiratory rate) collected from the subjects.
  All subjects who enrolled in this study (13 subjects in the placebo group and 12 subjects in the N RephasinⓇ SAL200 group) were defined as the Safety Set and included in the analysis.
Time Frame: up to 4 Week ± 5 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | N-Rephasin® SAL200
Number analyzed (Participants) | 13 | 12
Participants
  TEAE (Treatment-emergent AEs) | 12 | 10
  SAE | 2 | 2
  AEs leading to premature termination | 1 | 2

2. Secondary Outcome: Efficacy Endpoints 1
Description: Number of Participants With Negative Result in the First Blood Culture
Time Frame: by day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | N-Rephasin® SAL200
Number analyzed (Participants) | 13 | 12
Participants | 5 | 6

3. Secondary Outcome: Efficacy Endpoint 2
Description: The Proportion (Percentage) of Subjects who Died of Staphylococcus aureus Bacteremia Within 14 Days of Bacteremia Diagnosis
Time Frame: by day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | N-Rephasin® SAL200
Number analyzed (Participants) | 13 | 12
Participants | 1 | 1

4. Secondary Outcome: Efficacy Endpoint 3
Description: Proportion (Percentage) of Treatment Failure Against Staphylococcus aureus Bacteremia by Day 14
Time Frame: by day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | N-Rephasin® SAL200
Number analyzed (Participants) | 13 | 12
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Up to 4 weeks +5 Days
Arm/Group | Placebo | N-Rephasin® SAL200
All-Cause Mortality (participants affected / at risk) | 2/13 | 2/12
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/12
Other Adverse Events (participants affected / at risk) | 12/13 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | N-Rephasin® SAL200 (N=12)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Acute infarction (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure, type 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | N-Rephasin® SAL200 (N=12)
Constipation (Gastrointestinal disorders) | 6 (6) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 1 (1) — General disorders and administration site conditions
Chills (General disorders) | 0 (0) | 2 (3) — General disorders and administration site conditions
Asthenia (General disorders) | 0 (0) | 1 (1) — General disorders and administration site conditions
Chest discomfort (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Disease progression (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Facial pain (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Oedema peripheral (General disorders) | 0 (0) | 1 (1) — General disorders and administration site conditions
Pain (General disorders) | 0 (0) | 1 (1) — General disorders and administration site conditions
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Asterixis (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (4) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penis disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment into this study was terminated by the Sponsor prior to completion for strategic reasons (to initiate clinical development abroad).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT03089697/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03089697/SAP_001.pdf